CLINICAL TRIAL: NCT02985411
Title: Harvest for Health in Older Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Auburn University (Other)
Responsible Party: Principal Investigator, Wendy Demark-Wahnefried, PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: site garden; R01CA201362-01A1 (NIH)
Record Dates: First submitted 2016-12-03; First posted 2016-12-07 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-06

CONDITIONS: Cancer Survivor

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Gardening Intervention (Active Comparator): Wait-listed, will receive the gardening intervention after a 1-year period
  Interventions: Behavioral: Immediate Gardening Intervention
- Delayed Gardening Intervention (Active Comparator): Individuals in this group will serve as their own control
  Interventions: Other: Delayed Gardening Intervention

INTERVENTIONS:
Behavioral: Immediate Gardening Intervention — Provided with supplies to plan/plant 3 vegetable gardens over the course of a year. Survivors will be paired with a master gardener from their local Cooperative Extension to help guide them and provide mentorship in vegetable gardening,
  Arms: Immediate Gardening Intervention
Other: Delayed Gardening Intervention — Subjects will be monitored for 1-year and will then receive the same vegetable gardening intervention as described under the Immediate Gardening Intervention
  Arms: Delayed Gardening Intervention

SUMMARY:
Gardening interventions yield a multitude of measurable benefits that are evaluable within the context of a clinical trial. Harvest for Health forges new inroads in the delivery of holistic interventions to high risk populations, in this case, older cancer survivors. Since the intervention banks on an existing organization's infrastructure, it can easily be disseminated nationwide. The next step is to prove efficacy - an essential step in contributing to the science in this area, and one which is crucial for future dissemination.

DETAILED DESCRIPTION:
There are roughly 15 million cancer survivors in the US, comprising 4% of the populace. The number of cancer survivors is skyrocketing due to a confluence of the following factors: 1) Americans are aging; 2) cancer is an age-related disease (>60% of cancer survivors are age 65+); and 3) improvements in early detection and treatment have resulted in many common cancers having 5-year cure rates that surpass 90%. Rising numbers of cancer survivors is good news, but over $130 billion annually is needed to address subjects long-term health and psychosocial needs.113 Compared to others, cancer survivors are at higher risk for other cancers, CVD, osteoporosis, and diabetes. Accelerated functional decline also is a major problem for cancer survivors, especially those who are older. Baker et al. found that compared to age-matched controls, cancer cases (n=45,494) had significantly lower physical and social functioning, vitality, mental health, and HRQoL (p<0.001). Results of others are similar and suggest that cancer survivors face functional decline that threatens subject ability to live independently, posing a burden to themselves, subject families and the health care system. Programs exist in land grant universities in all 50 United States. Certified MGs complete > 100 hrs. of training and community service (CS) and 25 hrs./year of CS to maintain active status. In surveying 184 MGs in AL, the investigators found that 71% were "extremely interested" in mentoring a cancer survivor on vegetable gardening for subject CS, and an extra 26% stated that "they were interested and wanted to learn more." Thus, the project is of great interest and builds on an extant infrastructure for sustainability. Ultimately, this intervention could be disseminated to states with 3 growing seasons and adapted to colder weather in those with 2 growing seasons (36 states where 10.8 million older cancer survivors reside). The intervention also could be adapted for persons with other chronic diseases in which physical functioning and lifestyle behaviors are key. Finally, this project is significant because the intervention has great potential for sustainability since gardening: (a) involves many activities which prevent burn-out common with other forms of exercise, and allows participants to pursue PA outdoors which is related to greater enjoyment; (b) provides a sense of achievement and zest for life that come from nurturing and observing new life and growth; and (c) imparts natural prompts since plants require regular care (watering) and attention (harvesting) and serve as continual and dynamic behavioral cues.

ELIGIBILITY:
Inclusion Criteria:

* Residence in the following counties in Alabama: Autauga, Baldwin, Blount, Calhoun, Cherokee, Chilton, Coffee, Cullman, Dale, Dekalb, Elmore, Etowah. Houston, Jackson, Jefferson, Lauderdale, Lee, Limestone, Madison, Marshall, Mobile, Morgan, Montgomery, Pike, Randolph, Shelby, St. Clair, Tallapoosa, Tuscaloosa, Walker
* Diagnosed with one of the following cancers and completed primary treatment: localized larynx, gastric cardia, or cervix; localized or regionally-staged bladder, colorectum, fallopian tube, breast (female only), kidney and renal, melanoma, oral cavity, ovary, pharynx, prostate, soft tissue sarcoma, thyroid or uterus; or all stages: Hodgkin or Non-Hodgkin Lymphoma, Leukemia (CML CLL ALL) or testis.
* has at least one physical function limitation as measured by the SF-36 physical function subscale.

Exclusion Criteria:

* Currently tends an in-ground vegetable garden year round.
* Currently eats at least 2.5 cups of fruits and vegetable/day
* Currently obtains 150 or more of moderate-to-vigorous exercise per week
* Has a medical condition that precludes safe pursuit of gardening, i.e., severe orthopedic conditions, pending hip/knee replacement (within 6 mo.), paralysis, dementia, blindness, untreated stage 3 hypertension, or myocardial infarction, congestive heart failure, or conditions that required oxygen or hospitalization within 6 mo.
* unsuitable residence for gardening, i.e., no running water, inadequate sunshine.
* not able to speak or read English

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Percent of subjects in each group at year 1 who meet ALL 3 of 3 of the following goals: Physical performance tests, plasma α-carotene, and accelerometry-measured physical exam | 1 year after baseline
  Percent of subjects in each group at year 1 who meet ALL 3 of 3 of the following goals: Physical performance tests, plasma α-carotene, and accelerometry-measured PA
  * >5-point increase on the Short Form 36 Physical Function subscale [SF36 PFSS] AND improvement on the Senior Fitness Battery
  * Increase in intake of ½ c of vegetables and fruits/day AND increase is plasma alpha-carotene.
  * Increase of >30 minutes per week of moderate to vigorous physical activity AND confirmatory increase in physical activity as assessed by accelerometry.

SECONDARY OUTCOMES:
Mean Physical Functioning (SF36 physical function subscale) score in each group | 1 years after baseline
  The 10-item scale measures perceived limitations to various physical tasks in which the participant response "limited a lot," "limited a little" or "not limited at all" (A 3-point scale is used and the score is transformed to a 0-100 point scale in which a score of 50 reflects an average score (with a 100 reflecting no limitations and 0 means severe limitations in multiple domains
Mean physical performance (senior fitness battery) score | 1 year after baseline
  The Senior Fitness Test Battery tests several physical function domains: i.e., lower and upper body strength (using the 30-second chair stand and arm curl), endurance (using the 2-minute step test), flexibility (using the chair sit-and-reach and back scratch), and agility/dynamic balance (using the 8-ft Get Up & Go). Each test is backed by age and gender appropriate population-based norms; cutpoints denoting high risk for low function are as follows:
  * 30-second chair stand: <8 unassisted stands
  * Arm curl: <11 curls
  * 2-minute step test: <65 steps
  * Chair sit-and-reach: -4 cm in men and -2 cm in women
  * Back scratch: -4 cm in men and -2 cm in women
  * 8 foot Get up and Go: > 9 seconds
Mean vegetable and Fruit Consumption in each group | 1 year after baseline
  The number of daily ½ cup servings of vegetables and fruits will be measured by the Eating at America's Table Screener (EATS) questionnaire; this 10-item NCI-developed questionnaire will be able to assess whether individuals meet the goal (2.5 cups per day) or not.
Mean plasma alpha carotene value in each group | 1 year after baseline
  Plasma α-carotene will be quantified via high-performance liquid chromatography methods using a Hitachi 911clinical analyzer with standard chemistries by Roche (Indianapolis, IN). The range of α-Carotene varies from 0.1 to 0.90 μmol/ with a mean score of 0.5. This test is conducted for research purposes only. Thus, while a range between 0.50 and 0.90 is desirable, there are no clinically agreed guidelines to provide patients with information on lower levels.
Mean rate of physical activity (self report via the CHAMPS and accelerometry | 1 year after baseline
  Physical activity will be measured via self-report, using the Community Healthy Activities Models Program for Seniors (CHAMPS), a validated and sensitive tool that captures physical activities specific to older adults. This instrument will be used to assess minutes of moderate to vigorous activity per week. Objective levels of physical activity, will be captured via accelerometry. All participants will be asked to wear an activity monitor on their waist for 7 days at baseline, 1- and 2- year follow-up. Readings obtained from accelerometry also will be used to assess the minutes of moderate to vigorous physical activity.
Mean percent improvement on the Senior Fitness Battery test | 1 year post baseline
  Change from baseline to 1-year follow-up in each measure of physical performance will be compared between those in the immediate vs. delayed intervention groups at 1-year.
Mean percentage BMI score at 2 years post baseline | baseline to 2 years
  An improved diet and improved physical activity is associated with a weight status within the normal range, we will assess changes in weight status over the study period by measuring height (at baseline), and weight (using a platform scale) at all timepoints. Weights and heights will be converted to MI (KG/M2). The percentage of each study arm categorized as normal weight (BMI 18.5 - 24.9) at each time point.
Mean Quality of Life (SF36) score at 2 years | 2 years after baseline
  The SF-36 offers scores for mental health and physical health. These scores are each transformed to a 0-100 point scale in which a score of 50 reflects an average score (with a 100 reflecting optimal status and 0 meaning severly compromised (minimal) status
Mean telomerase score in each group | 1 year post baseline
  PENDING RECEIPT OF ANCILLARY FUNDING: Telomerase activity will be measured in blood sample buffy coats using the Telomerase PCR ELISA assay (Boehringer Mannheim). While many individuals will express non-detectable levels, the percentage of individuals who have optimal levels of 0.20-1.5 will be compared in each arm
Mean IL-6 and TNF alpha score in each arm | 1 year post baseline
  IL-6 will be assessed IN PLASMA via electrochemiluminescence (Meso-scale Discovery; Gaithersburg, MD). AN ANTICIPATED RANGE OF 0.015 to 11.5 pg/ml IS ANTICIPATED, WITH LOWER LEVELS INDICATING LESS INFLAMMATION AND LOWER RISK FOR CHRONIC DISEASE (VALUES <1.47)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Demark-Wahnefried, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Will not share data until study is complete and all data deidentified

REFERENCES:
- [Background] Cases MG, Fruge AD, De Los Santos JF, Locher JL, Cantor AB, Smith KP, Glover TA, Cohen HJ, Daniel M, Morrow CD, Moellering DR, Demark-Wahnefried W. Detailed methods of two home-based vegetable gardening intervention trials to improve diet, physical activity, and quality of life in two different populations of cancer survivors. Contemp Clin Trials. 2016 Sep;50:201-12. doi: 10.1016/j.cct.2016.08.014. Epub 2016 Aug 23. PMID 27565830
- [Background] Blair CK, Madan-Swain A, Locher JL, Desmond RA, de Los Santos J, Affuso O, Glover T, Smith K, Carley J, Lipsitz M, Sharma A, Krontiras H, Cantor A, Demark-Wahnefried W. Harvest for health gardening intervention feasibility study in cancer survivors. Acta Oncol. 2013 Aug;52(6):1110-8. doi: 10.3109/0284186X.2013.770165. Epub 2013 Feb 26. PMID 23438359
- [Background] Demark-Wahnefried W, Cases MG, Cantor AB, Fruge AD, Smith KP, Locher J, Cohen HJ, Tsuruta Y, Daniel M, Kala R, De Los Santos JF. Pilot Randomized Controlled Trial of a Home Vegetable Gardening Intervention among Older Cancer Survivors Shows Feasibility, Satisfaction, and Promise in Improving Vegetable and Fruit Consumption, Reassurance of Worth, and the Trajectory of Central Adiposity. J Acad Nutr Diet. 2018 Apr;118(4):689-704. doi: 10.1016/j.jand.2017.11.001. Epub 2018 Jan 2. PMID 29305129
- [Background] Bail JR, Fruge AD, Cases MG, De Los Santos JF, Locher JL, Smith KP, Cantor AB, Cohen HJ, Demark-Wahnefried W. A home-based mentored vegetable gardening intervention demonstrates feasibility and improvements in physical activity and performance among breast cancer survivors. Cancer. 2018 Aug;124(16):3427-3435. doi: 10.1002/cncr.31559. Epub 2018 Jun 22. PMID 29932460
- [Derived] Demark-Wahnefried W, Oster RA, Smith KP, Kaur H, Fruge AD, Cole WW, Locher JL, Rocque GB, Pisu M, Bail JR, Cohen HJ, Moellering DR, Blair CK. Vegetable Gardening and Health Outcomes in Older Cancer Survivors: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2417122. doi: 10.1001/jamanetworkopen.2024.17122. PMID 38900426
- [Derived] Bail JR, Blair CK, Smith KP, Oster RA, Kaur H, Locher JL, Fruge AD, Rocque G, Pisu M, Cohen HJ, Demark-Wahnefried W. Harvest for Health, a Randomized Controlled Trial Testing a Home-Based, Vegetable Gardening Intervention Among Older Cancer Survivors Across Alabama: An Analysis of Accrual and Modifications Made in Intervention Delivery and Assessment During COVID-19. J Acad Nutr Diet. 2022 Sep;122(9):1629-1643. doi: 10.1016/j.jand.2022.05.005. Epub 2022 May 6. PMID 35533876
- [Derived] Kaur H, Fernandez JR, Locher JL, Demark-Wahnefried W. Rural and Urban Differences in Vegetable and Fruit Consumption Among Older Cancer Survivors in the Deep South: An Exploratory Cross-Sectional Study. J Acad Nutr Diet. 2022 Sep;122(9):1717-1724.e4. doi: 10.1016/j.jand.2022.01.003. Epub 2022 Jan 10. PMID 35017097
- [Derived] Warnock AC, Kaur H, Buckman JR, Hoenemeyer T, Demark-Wahnefried W. A comparison of two mail-based strategies to recruit older cancer survivors into a randomized controlled trial of a lifestyle intervention. J Cancer Surviv. 2022 Oct;16(5):998-1003. doi: 10.1007/s11764-021-01091-x. Epub 2021 Aug 3. PMID 34342814